CLINICAL TRIAL: NCT06927258
Title: Application of Changyanning Granule in Endoscopic Resection of Colorectal Polyps
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0661
Record Dates: First submitted 2024-10-18; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Polyps
Keywords: colorectal polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Changyanning group (Active Comparator): The Changyanning group takes Changyanning granules starting from 1 day before surgery until 5 days after surgery. The granules are taken preoperatively at the same time as the first dose of laxative, and postoperatively starting after resuming an open diet.
  Interventions: Drug: changyanning granules
- The control group (Placebo Comparator): The control group does not use Changyanning granules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: changyanning granules — From one day before the procedure to five days postoperatively, patients in the experimental group will be administered Chanyanning granules.
  Other Names: control
  Arms: The Changyanning group
Drug: Placebo — control
  Arms: The control group

SUMMARY:
This study aims to evaluate the efficacy of Chanyanning granules in patients undergoing endoscopic resection of colorectal polyps with a basal diameter of 5-30 mm. From one day before the procedure to five days postoperatively, patients will be administered Chanyanning granules. The study will observe intraoperative and postoperative bleeding, perforation, and digestive system-related clinical symptoms such as postoperative abdominal pain, bloating, diarrhea, constipation, hematochezia, and fatigue, as well as related inflammatory markers, to determine the therapeutic effect of Chanyanning granules.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colorectal polyps through endoscopic examination and who received corresponding endoscopic treatments (EMR, hybrid ESD, ESD).

Exclusion Criteria:

* Concurrent infectious diseases or malignant tumors; Accompanied by severe cardiopulmonary diseases (such as severe heart failure, COPD, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
serum interleukin-6 | From enrollment to the end of treatment at 2 weeks
The incidence of complications | From enrollment to the end of treatment at 2 weeks
  The incidence of complications (blood in stool, perforation) and postoperative discomfort symptoms (abdominal pain, abdominal distension, diarrhea, constipation, fatigue, fever, etc.) were compared between the experimental group and the control group (primary endpoints).
white blood cells | From enrollment to the end of treatment at 2 weeks
C-reactive protein | From enrollment to the end of treatment at 2 weeks
erythrocyte sedimentation rate | From enrollment to the end of treatment at 2 weeks

SECONDARY OUTCOMES:
hospital stay | From enrollment to the end of treatment at 2 weeks
hospitalization costs | From enrollment to the end of treatment at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China